CLINICAL TRIAL: NCT06823908
Title: in Vitro Evaluation of the Anti-fibrotic Activity of Adipose Tissu-derived Stromal Vascular Fraction Used as a Medicinal Treatment for Scarred Vocal Folds: Interest in the Definition of 'Potency' Markers and Optimized Cellular Engineering Trategies
Brief Title: in Vitro Evaluation of the Anti-fibrotic Activity of Adipose Tissu-derived Stromal Vascular Fraction Used as a Medicinal Treatment for Scarred Vocal Folds
Acronym: CELLCORDES BIO
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Collaborators: Aix Marseille Université (Other)
Responsible Party: Sponsor
Other Study IDs: RCAPHM24_0513
Record Dates: First submitted 2025-02-07; First posted 2025-02-12 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-04

CONDITIONS: Vocal Cord Injuries

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- heathly donors: patients who come as part of their routine care
  Interventions: Other: Reuse of surgical waste
- CELLCORDES 2 Patient: Patient included in the clinical trial CELLCORDES 2
  Interventions: Other: Reuse of biological samples

INTERVENTIONS:
Other: Reuse of surgical waste — Heathly donnors will be received in the plastic surgery department as part of routine care. They will be informed of the study and their surgical waste (adipose tissue) will be recovered specifically for this research.
  Groups: heathly donors
Other: Reuse of biological samples — Patients included in the cellcordes 2 trial who have given their consent for the re-use of their biological samples (Stromal Vascular Fraction) in other clinical research projects, and who have been informed of the cellcordes bio study.
  Groups: CELLCORDES 2 Patient

SUMMARY:
This is a single-center, prospective study, aimed at investigating the anti-fibrotic in vitro activity of the stromal vascular fraction of patients with scarred vocal cord.

DETAILED DESCRIPTION:
This single-center, prospective study will last 28 months and will be carried out in two stages:

1. Comparison of the in vitro anti-fibrotic activity and production/management circuit of different cell therapy products derived from adipose tissue obtained from healthy donors (n=8) [secondary objective] during the first 12 months of the project.
2. Evaluate the association between the in vitro anti-fibrotic activity of fraction vascular fraction (FVS) samples and the clinical improvement obtained with the same sample autologously injected into a patient in the CELLCORDES2 trial (minimum recruitment n=10, CELLCORDES2 biocollection) [primary objective]. This second stage will be carried out between M12 and M24 to optimize the number of patients to be included.

ELIGIBILITY:
Inclusion criteria for patients included in the CELLCORDES 2 clinical trial

* Voice Handicap Index > 50/120
* Scarring, congenital (sulcus) or post-phonosurgery vocal cords
* Vibratory anomalies in the middle third of one or both vocal cords on stroboscopy
* A minimum of six months after the initial surgery
* Patients aged 18 to 70 years
* Good general health
* Negative pregnancy test and contraception for women of childbearing age Signature of consent for the storage and use of biological samples

Inclusion criteria for Healthy donnors:

* Liposuction surgery for aesthetic reasons
* BMI between 18 and 27
* No chronic diseases
* Non-opposition to the use of surgical waste for research purposes after freezing in a biological collection

Exclusion criteria: For all patients:

* Refusal or inability to comply with the study procedures
* Minors
* Pregnant or breastfeeding women
* Legally protected adults (under guardianship or curatorship)
* Individuals residing in a healthcare or social establishment emergency situations
* Individuals deprived of liberty
* Detainees
* Individuals not covered by a social security scheme
* Use of an experimental drug in the last three months
* Contraindication to local anesthesia
* Anticoagulant treatment
* Coagulation disorders (TP < 65%, TCA > 1.2)
* Premenopausal women of childbearing age without contraception
* Lack of or refusal of informed consent

Exclusion criteria for Patients in the CELLCORDES 2 clinical trial:

* Patients refusing pre- and post-operative speech therapy
* History of malignant lesions or severe dysplasia on the scarred vocal cord
* History of laryngeal papillomatosis
* Active infectious diseases
* Positive serology for HIV1 and 2, p24 Ag, HCV Abs, HBs Ag, HbC Abs, HTLV and II Abs, TPHA
* Need for perioperative antibiotic prophylaxi

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with scared vocal cord
Sampling Method: Non-Probability Sample
Enrollment: 18 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-04 (Estimated); Study Completion 2027-10 (Estimated)

PRIMARY OUTCOMES:
collagene protein levels | 24 months
  The stromal vascular fraction of patient will be co-cultured with an in-vitro model of scarred vocal cord. Then, the levels of collagene will be quantified by western blot to measure the anti-fibrotic activity of SVF.
Actine alpha 2 (ACTA2) RNA levels | 24 months
  The stromal vascular fraction of patient will be co-cultured with an in-vitro model of scarred vocal cord. Then, the levels of ACTA2 will be quantified by RT-qPCR to measure the anti-fibrotic activity of SVF.
Alpha Smooth muscle actin (aSMA) protein levels | 24 months
  The stromal vascular fraction of patient will be co-cultured with an in-vitro model of scarred vocal cord. Then, the levels of aSMA will be quantified by western blot to measure the anti-fibrotic activity of SVF.
collagen type 1 alpha 1 chain (COL1A1) RNA levels | 24 months
  The stromal vascular fraction of patient will be co-cultured with an in-vitro model of scarred vocal cord. Then, the levels of COL1A1will be quantified by RT-qPCR to measure the anti-fibrotic activity of SVF.

SECONDARY OUTCOMES:
collagene protein levels | 24 months
  Cellular products obtained from adipose tissue obtained from healthy donnors will be co-cultured with an in-vitro model of scarred vocal cord. Then, the levels of collagen will be quantified by western blot to measure the anti-fibrotic activity of different cellular products.
Actine alpha 2 (ACTA2) levels | 24 months
  Cellular products obtained from adipose tissue of healthy donnors will be co-cultured with an in-vitro model of scarred vocal cord. Then, the levels of ACTA2 will be quantified by RT-qPCR to measure the anti-fibrotic activity of different cellular products.
Alpha Smooth muscle actin (aSMA) protein levels | 24 months
  Cellular products obtained from adipose tissue of healthy donnors will be co-cultured with an in-vitro model of scarred vocal cord. Then, the RNA levels of aSMA will be quantified by western blot to measure the anti-fibrotic activity of different cellular products
ollagen type 1 alpha 1 chain (COL1A1) RNA levels | 24 months
  Cellular products obtained from adipose tissue of healthy donnors will be co-cultured with an in-vitro model of scarred vocal cord. Then, the RNA levels of COL1A1 will be quantified by RT-qPCR to measure the anti-fibrotic activity of different cellular products.

CONTACTS AND LOCATIONS:
Overall Officials: MATTEI Alexia, Doctor, Principal Investigator — assistance publique - hôpitaux de Marseille

IPD SHARING:
Plan to Share IPD: Undecided